CLINICAL TRIAL: NCT03467789
Title: Vitamin D as a Nutritional Neoadjuvant During Photodynamic Therapy of Basal Cell Carcinoma in Basal Cell Nevus Syndrome
Brief Title: Vitamin D as a Nutritional Neoadjuvant During Photodynamic Therapy of Basal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CASE5617; NCT03483441 (obsolete NCT alias)
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Basal Cell Carcinoma; Basal Cell Nevus Syndrome
Keywords: Vitamin D; Photodynamic Therapy
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: Each patient serves as his/her own control. Two PDT sessions are given, constituting Arm 1 and Arm 2. Arm 1 is placebo pill, then PDT. Arm 2 is Vit D pill, then PDT. In any given patient, the order of Arm 1 vs. Arm 2 will be randomized.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither the participant nor the treating physicians will know which patients receive the Vitamin D3 or placebo pills. Using a "coin toss" approach, the Research Pharmacist will assign each patient to a study group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: D3 prior to first PDT (Experimental): In both groups, one PDT session is preceded by neoadjuvant PDT while the other PDT session has no pretreatment.
  Group A will take dietary D3 pills prior to the first PDT treatment (day 1), and placebo pills prior to the second PDT treatment (at 2 months). Both Group A and Group B will take continuous serum D3 prior to the third PDT visit (Month 4). A final assessment of lesion clearance will be performed at 6 months
  Interventions: Drug: Dietary Vitamin D3 pre-treatment; Radiation: Photodynamic therapy; Drug: Serum Maintenance Vitamin D3
- Group B: D3 prior to second PDT visit (Experimental): In both groups, one PDT session is preceded by neoadjuvant PDT while the other PDT session has no pretreatment.
  Group B will receive placebo prior to their first PDT visit (day 1), and Vitamin D3 prior to their second PDT visit (at 2 months). Both Group A and Group B will take continuous D3 prior to the third PDT visit (Month 4). A final assessment of lesion clearance will be performed at 6 months
  Interventions: Drug: Dietary Vitamin D3 pre-treatment; Radiation: Photodynamic therapy; Drug: Serum Maintenance Vitamin D3

INTERVENTIONS:
Drug: Dietary Vitamin D3 pre-treatment — The daily dose of D3 will always be 10,000 IU/day. Total amounts of D3 supplementation given will be adjusted, based upon serum 25-hydroxy-D3 levels found at baseline. Duration of pretreatment will be 14 days if the D3 level is < 31 ng/mL, and 5 days if the D3 level is > 31 ng/mL
Radiation: Photodynamic therapy — Photodynamic Therapy (PDT) is an experimental technique that works by combining a photosensitizing topical agent and an intense light source to kill tumor cells.
  Other Names: PDT
Drug: Serum Maintenance Vitamin D3 — 2,000 IU/d for adults, 1,000 IU/d for children taken after third visit.

SUMMARY:
The purpose of this study is to study 50 patients with multiple Basal Cell Carcinoma (BCC) who will be receiving Photodynamic Therapy (PDT) as treatment for their tumors. This study wants to establish the optimal conditions for treating BCC tumors with PDT. Previous research suggests that taking Vitamin D prior to the start of PDT could help improve the effectiveness of the treatment in eliminating the BCC. Overall, this study will help establish oral Vitamin D3/PDT as a new combination therapy for skin cancer (BCC).

Photodynamic Therapy (PDT) is an investigational (experimental) technique that works by combining a photosensitizing topical agent and an intense light source to kill tumor cells. PDT is currently approved for the treatment of BCC in Europe, Canada, and Australia. However, it is experimental in the United States because it is not approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The overall hypothesis is that PDT could provide exceptional benefit in patients with Basal Cell Nevus Syndrome (BCNS) and multiple BCC tumors because PDT is nonmutagenic, nonscarring, and can be safely repeated many times. The specific study hypothesis is that Vitamin D might be useful as a neoadjuvant to improve tumor responses to PDT. In preclinical studies, the investigators showed that epithelial tumors are more responsive to aminolevulinic acid (ALA)-based PDT when "primed" by pre-exposure to the dietary form of Vitamin D (cholecalciferol, D3). This study will test the hypothesis that oral D3 supplements, administered over a relatively short time, can boost the effectiveness of PDT for cutaneous (BCC) in this patient population. Patients with BCNS and multiple BCC, or normal patients with at least 3 BCC tumors, will be enrolled. They will receive three PDT treatments, at two-month intervals, over a 6 month period.

Primary Objective

• To determine tumor clinical clearance rates after neoadjuvant D3/PDT, and after PDT alone. To accomplish this, the first two PDT treatments in each study patient will be randomized, i.e. one PDT session will be performed after D3 pretreatment, the other without any pretreatment.

Secondary Objective(s)

* To assess the level of PpIX accumulation in BCC lesions at various treatment visits, in the absence or presence of neoadjuvant D3. (Fluorescence dosimetry measurements)
* To assess tolerability of the technique. (Pain scale measurements)
* To assess patient satisfaction with the technique. (Cosmetic result, and questionnaire)
* To assess D3 serum levels (in serum) and VDR status (in leukocyte DNA), and correlate these results to clinical outcomes.

Study Design:

In this clinical study, each patient will serve as his or her own control with respect to BCC tumor responsiveness to neoadjuvant D3 supplementation. The first two PDT treatments will be randomized. Thus, patients in Group A will take D3 pills prior to the first PDT treatment, and placebo pills prior to the second PDT treatment. For patients in Group B, the order is reversed. Total amounts of D3 supplementation given will be adjusted, based upon serum 25-hydroxy-D3 levels found at baseline. Patients with VD deficiency will take 14 days of neoadjuvant D3, vs. only 5 days if the initial VD level is normal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Basal Cell Nevus Syndrome (BCNS) as defined in the Consensus Statement from the first International colloquium on BCNS.

  * Major Criteria are:

    * (1) BCC prior to age 20 years, or excessive number of BCCs out of proportion to prior sun exposure and skin type;
    * (2) keratocyst of the jaw prior to age 20;
    * (3) palmar or plantar pitting;
    * (4) lamellar calcification of the falx cerebri;
    * (5) medulloblastoma;
    * (6) first degree relative with BCNS;
    * (7) Patched-1 (PTCH1) gene mutation.
  * Minor Criteria are:

    * (1) rib anomalies, or other specific skeletal malformations including kyphoscoliosis and short 4th metacarpals;
    * (2) macrocephaly;
    * (3) cleft/lip or palate;
    * (4) fibroma of the heart or ovary;
    * (5) ocular abnormalities;
  * For diagnosis of BCNS, the participant must have either 2 major criteria, one major and two minor criteria.
* At least three BCC tumors, two of which are biopsy-proven
* Female subjects must not become pregnant during the study
* Subjects must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Pregnant or nursing.
* At risk for hypercalcemia (renal disease, sarcoidosis, etc.)
* Taking vismodegib or a hedgehog pathway inhibitor; must stop at least 3 months prior to visit 1.
* Taking any topical treatment on their BCC tumors; must stop at least 1 month prior.
* Taking Vitamin D or multivitamin supplements; must stop at least 1 month prior.
* Currently undergoing treatment for other cancers with medical or radiation therapy.
* Participants with a known hypersensitivity to 5-aminolevulinic acid or any component of the study material.
* Participants with history of a photosensitivity disease, such as porphyria cutanea tarda.
* Currently participating in another clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
BCC: Rate of tumor clearance | Up to 6 months after first treatment visit
  Change in tumor diameter per month. For each participant, the investigators will analyze the difference in tumor clearance between treatments, one with neoadjuvant D3+PDT, the other with PDT alone, and the other with or without D3 in order to establish a D3 replete state. The order of the first two treatments is randomized in case the assumption of a linear tumor clearance rate is incorrect
  The statistical significance of the difference in Delta-T after D3+PDT versus the difference in Delta-T after PDT alone will be tested using ANOVA.

SECONDARY OUTCOMES:
BCC: Level of protoporphyrin IX (PpIX) accumulation in BCC lesions | Up to 6 months after first treatment visit
  For each patient, whether in the absence or presence of neoadjuvant Vitamin D3, assessments of PpIX accumulation in BCC lesions using fluorescence dosimetry measurements will be made at selected treatment visits.
Serum 25-hydroxy-vitamin D3 (25OH-D3) levels | Up to 6 months after first treatment visit
  Using a 10mL blood sample, a 25OH-D3 assay will be used to determine D3 levels in the blood
Number of patients with active form of leukocyte DNA vitamin D Receptor (VDR) | Up to 6 months after first treatment visit
  Study team will collect patients' leukocyte DNA and examine the VDR gene sequences directly. Patients with the active VDR allele are postulated to have better PDT outcomes
Pain scale measurement | Up to 6 months after first treatment visit
  average pain scale measurements to assess tolerability of the technique to be taken in the week following each PDT treatment (3 total). Ranging from 0 to 10 where 0 indicates no pain and 10 indicates the worst pain possible
Erythema score | Up to 6 months after first treatment visit
  A measure of Patient Satisfaction Score. Score from photographs on a scale from 1-4 with higher scores indicating more erythema
Satisfaction with treatment outcome from the technique | Up to 6 months after first treatment visit
  A participant satisfaction questionnaire will be administered at the final study visit measuring the participant's satisfaction with the treatment outcome on a 5 point scale (Extremely Satisfied to Extremely Dissatisfied)
Satisfaction with cosmetic outcome from the technique | Up to 6 months after first treatment visit
  A participant satisfaction questionnaire will be administered at the final study visit measuring the participant's satisfaction with the cosmetic outcome on a 5 point scale (Extremely Satisfied to Extremely Dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Edward V. Maytin, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio